CLINICAL TRIAL: NCT07111455
Title: Prospective Cohort Study on Oral Microbiome Changes in Patients With Locally Advanced Oral Squamous Cell Carcinoma Following Neoadjuvant Chemoimmunotherapy
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-KY-189
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Oral Squamous Cell Carcinoma
Keywords: Oral Microbiome; Neoadjuvant Chemoimmunotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 16S rRNA Swab Sample from Oral Tumor;Saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exposed Group: Participants were planned to receive 2 cycles of intravenous neoad- juvant Tislelizumab (200 mg) every 3 weeks,and Paclitaxel 135-175mg/m² ,Cisplatin 80-120mg/m² or Carboplatin 0.3-0.4g/m² through intravenous infusion each 3-week cycle for 2 cycles.

SUMMARY:
Investigating the Relationship Between Oral Microbiome Alterations and Tumor Markers in Locally Advanced Oral Squamous Cell Carcinoma (LA-OSCC) After Neoadjuvant Chemoimmunotherapy: Implications for Therapeutic Efficacy, Chemoresistance, and Prognostic Assessment

ELIGIBILITY:
Inclusion Criteria:

1. Oral squamous cell carcinoma (OSCC) diagnosed as locally advanced (T3N0M0, T1-3N1M0, T4aN0-2M0, T1-4aN3M0, or T4bN0-3M0) according to AJCC staging criteria.
2. Their age ranged from 18 to 80 years;regardless of gender.
3. Absence of prior head and neck radiation therapy or chemotherapy.
4. Adequate blood function: white blood cell count (WBC) >＝3.5×10^9/L, platelet count (PLT) >＝75×10^9/L：Hemoglobin concentration (HGB) >＝90g/L.
5. Adequate liver function： total bilirubin (TBIL) <＝ the upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <＝2.5 times the upper limit of normal.
6. Adequate renal function：estimated glomerular filtration rate (eGFR) greater than 45 mL/min per 1.73 m².
7. The heart, brain, lung and other vital organs function and general condition can tolerate NACI.
8. PS score <＝2.
9. Signed informed consent form and voluntarily agreeing to participate in this study.

Exclusion Criteria:

1. Pregnancy or lactation (for female participants).
2. Patients with a history of epilepsy or psychiatric disorders that were not well-controlled.
3. Patients with severe allergic diathesis or suspected or confirmed alcohol or drug addiction.
4. Patients who had taken antibiotics within 7 days before enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced oral squamous cell carcinoma (OSCC) attending the Department of Stomatology, Zhujiang Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 8 weeks
  According to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, it is defined as the proportion of patients who achieved Complete Response (CR) or Partial Response (PR).Complete Response (CR) was defined as disappearance of all target lesions. Partial Response (PR) was defined as >=30% decrease in the sum of the longest diameter of target lesions.

SECONDARY OUTCOMES:
two-year overall survival rate | 24 months
  The proportion of patients surviving ≥2 years post-treatment
two-year progression-free survival rate | 24 months
  The proportion of patients who remain alive and progression-free for 2 years after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Stomatology, Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No